CLINICAL TRIAL: NCT01720264
Title: A Multicenter Phase II Trial of Inhibition of CD26 Peptidase Using Sitagliptin to Enhance Engraftment After Umbilical Cord Blood Transplantation for Adults With Hematological Malignancies
Brief Title: Multicenter Phase II of CD26 Using Sitagliptin for Engraftment After UBC Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sherif S. Farag (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Sherif S. Farag, Lawrence H. Einhorn Professor of Oncology, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1208009261; HL112669; 1R01HL112669-01 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-02 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Hematopoetic Myelodysplasia; Leukemia, Myelogenous, Chronic; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sitagliptin (Experimental): Sitagliptin q 12 hours PO starting on Day -1 then given every 12 hours (total 10 doses) on Day 0, Day +1, +2 and Day +3.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin q 12 hours PO starting on Day -1 then given every 12 hours (total 10 doses) on Day 0, Day +1, +2 and Day +3.
  Other Names: Januvia

SUMMARY:
The main purpose of this trial is to assess the efficacy and safety of sitagliptin in enhancing engraftment following umbilical cord blood transplantation (recovery of blood counts after transplant).

DETAILED DESCRIPTION:
Umbilical cord blood (UCB) is more commonly used for transplantation in children but is being used in adults more often. However, because adults are larger than children, the relatively smaller stem cell dose in UCB is major limitation for transplantation in adults and engraftment can be delayed. This study is trying to find out if the drug sitagliptin can be used to increase and speed up engraftment in adults receiving UCB transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following disease types:

  * Acute myeloid leukemia (AML) with disease features as described in the protocol.
  * Acute lymphoblastic leukemia (ALL) with disease features as described in the protocol.
  * Myelodysplasia with disease features as described in the protocol.
  * Chronic myelogenous leukemia (CML) with disease features as described in the protocol.
  * Patients with aggressive non-Hodgkin's lymphoma (NHL), including diffuse large cell lymphoma, mediastinal B-cell lymphoma, transformed lymphoma, mantle cell lymphoma, and peripheral T cell lymphoma, who also have one of the disease features as described in the protocol.
* At least 35 days following start of preceding leukemia induction cytotoxic chemotherapy.
* For patients in remission, there should be no readily available consenting HLA-matched related donor who is either matched fully matched or mismatched at only one locus of HLA-A, -B, and DRB1.
* No availability of a readily available HLA-matched volunteer unrelated donor (8 of 8 allele match at HLA-A, -B, -C and -DRB1).
* Patients must have a matched or partially matched UCB unit with >/= 2.5 x10^7 nucleated cells/kg of recipient weight at the time of cryopreservation.
* No current uncontrolled bacterial, viral or fungal infection (defined as currently taking medication and progression of clinical symptoms).
* No HIV disease.
* Non pregnant and non-nursing.
* Required baseline laboratory values as described in the protocol.
* Signed written informed consent.

Exclusion Criteria:

* Symptomatic uncontrolled coronary artery disease or congestive heart failure.
* Severe hypoxemia with room air PaO2<70, supplemental oxygen dependence, or DLCO<50% predicted.
* Patients with central nervous system (CNS) involvement refractory to intrathecal chemotherapy.
* Prior allogeneic or autologous hematopoietic stem cell transplant in the last 6 months.
* Patients who are taking other insulin secretagogues and/or insulin.
* Patients who have hypersensitivity to sitagliptin.
* Patients with a history of pancreatitis, cholelithiasis, alcoholism, or fasting hypertriglyceridemia (> 2 x ULN).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2016-08-27 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif S Farag, MBBS, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - New York Medical College/Westchester Medical Center/Maria Fareri Children's Hosptial, Valhalla, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was stopped at 15 patients due to poor accrual. One patient subsequently found not to have met eligibility because she commenced treatment one day earlier than the prescribed 35-day interval from previous therapy is included in the analysis.
Groups:
- Sitagliptin: Sitagliptin 600 mg q 12 hours PO for a total of 10 doses plus Total Body Irradiation (TBI) or Chemotherapy only.
Period: Transplant With Sitagliptin for 15 Days
Arm/Group | Sitagliptin
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1
Period: Post-transplant (Day 16) to 1 Year
Arm/Group | Sitagliptin
Started | 14
Completed | 2
Not Completed | 12
Not completed — Death | 8
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin: Sitagliptin 600 mg q 12 hours PO for a total of 10 doses plus Total Body Irradiation or Chemotherapy only.
Arm/Group | Sitagliptin
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (13.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Subjects Engrafting by Day +30 After Transplantation
Description: Percent of patients and the 95% Binomial Confidence interval who were able to achieve neutrophils engraftment (defined as the date of the first of three consecutive ANC values obtained on different days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l) by 30 days following transplant.
Time Frame: Day 0 to Day +30 post transplant
Population: All patients who received treatment and were followed after transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 15
percentage of participants | 100 [78 to 100]

2. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. Patients surviving at least 14 days after transplant will be evaluable for this endpoint. Patients who did not have neutrophil engraftment before death will be censored at the date of death. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients who received treatment and survived at least 14 days after transplant.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitagliptin
Number analyzed (Participants) | 15
days | 19 [13 to 20]

3. Secondary Outcome: Time to Platelet Engraftment
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of three consecutive Complete Blood Counts (CBCs) obtained on different days after transplantation during which the platelet count is at least 20 x109/l. The CBCs obtained should be at least seven days after the most recent platelet transfusion. Only patients who achieved engraftment of platelets will be included in the analysis. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) up to 1 year
Population: All patients who received treatment and who achieved platelet recovery/engraftment of platelets.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitagliptin
Number analyzed (Participants) | 6
days | 52 [21 to 89]

4. Secondary Outcome: Number of Subjects With Treatment Related Adverse Events Grade 3 and 4 Non-hematological Toxicities
Description: Number of unique patients who had a treatment related (possible, probable or definite) non-hematological adverse event that was graded 3 or greater.
Time Frame: Day 0 up to 3 years
Population: All patients enrolled and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=15)
Cardiac arrest (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 2
Hepatitis viral (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 3
Meningitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Capillary leak syndrome (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=15)
Anemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fever (General disorders) | 3
Localized edema (General disorders) | 2
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 2
Bladder infection (Infections and infestations) | 1
Encephalitis infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 10
Lung infection (Infections and infestations) | 2
Rhinitis infective (Infections and infestations) | 1
Salivary gland infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 6
Creatinine increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 3
Hydrocephalus (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Menorrhagia (Reproductive system and breast disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes